CLINICAL TRIAL: NCT02816086
Title: A New Interdisciplinary Collaboration Structure in Secondary and Primary Care to Improve Medication Safety in the Elderly
Brief Title: A New Interdisciplinary Collaboration Structure to Improve Medication Safety in the Elderly
Acronym: IMMENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016/41366
Record Dates: First submitted 2016-05-30; First posted 2016-06-28 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2020-08

CONDITIONS: Health Services for the Aged; Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): The study participants receives standard care in the ward, this does not include a pharmacist.
- Intervention (Experimental): Interdisciplinary collaboration structure
  Interventions: Other: Interdisciplinary collaboration structure

INTERVENTIONS:
Other: Interdisciplinary collaboration structure — A pharmacist is integrated in the team surrounding the patient, working by the Integrated Medicines Management (IMM) model. The IMM-model consist of medication reconciliation, medication review, standardized medication reports and counseling patients about their medication at discharge. In addition a phone meeting between the primary care physician and the study pharmacist is added after discharge.
  Arms: Intervention

SUMMARY:
Suboptimal use of medications among geriatric patients is well-known problem and leads to medication errors, re-hospitalizations and death. By using a randomized controlled trial (RCT) design the investigators aim to explore a new inter-professional working structure. The working structure is based on the scientifically and clinically acknowledged integrated medicines management (IMM) model. The overall aim of the study is to explore the effect of the new working structure on the composite endpoint re-hospitalization + visit to an emergency department during 12 months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥70 years
* Admitted to the geriatric internal medicine ward in the University Hospital of North Norway (UNN) Tromsø or the general internal medicine ward in UNN Harstad.
* Willing to provide written informed consent during hospital stay (patient or next of kin)

Exclusion Criteria:

* Unable to communicate in Norwegian (patient or next of kind)
* Terminally ill, e.g cancer in end-life stage
* Control group patients where the physician request an assessment from a pharmacist
* Time from admittance to the ward to inclusion is more than 72 hours
* Occupying a bed in the study wards but under the care of physicians from a non-study ward.
* Planned discharged on the inclusion day

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 516 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Emergency medical visits | 12 months after hospital discharge
  Rate of emergency Medical visits at 12 months. Emergency Medical visits is a composite endpoint including emergency department visits and unscheduled hospitalization

SECONDARY OUTCOMES:
Self-reported quality of life | 1 months after hospital discharge
  Change in self-reported quality of life using the validated EQ-5D
Self-reported quality of life | 6 months after hospital discharge
  Change in self-reported quality of life using the validated EQ-5D
Self-reported quality of life | 12 months after hospital discharge
  Change in self-reported quality of life using the validated EQ-5D
length in days of index hospital stay | Days from hospitalization to discharge of index hospital stay, assessed up to 12 months
  Days from hospital admission to discharge of index hospital stay
Time to first rehospitalization | First rehospitalization after discharge from index hospital stay, up to 12 months after discharge.
  Days to first hospitalization
Visits to primary care physician | 12 months after discharge for index hospital stay
  Visitation rate at 12 months
Mortality rate | 12 months after randomization
Total score of the Medication appropriateness index (MAI) | Baseline at randomization
Change in total score of the Medication appropriateness index (MAI) | From baseline to date of discharge from hospital, assessed up to 12 months
Inappropriate medications identified through the Norwegian general practice criteria (NORGEP) | Baseline at randomization
Change in Inappropriate medications identified through the Norwegian general practice criteria (NORGEP) | From baseline to date of discharge from hospital, assessed up to 12 months
Change in inappropriate medications identified through the Norwegian general practice criteria (NORGEP) | From baseline to 3 months after discharge from index hospital stay, assessed up to 12 months
Potentially inappropriate prescribing identified through the Screening Tool to Alert doctors to Right treatment (START) | Baseline at randomization
Change in potentially inappropriate prescribing identified through the Screening Tool to Alert doctors to Right treatment (START) | From baseline to date of discharge from hospital, assessed up to 12 months
Potentially inappropriate prescribing identified through the Screening Tool of Older Persons' Prescriptions (STOPP) | Baseline at randomization
Change in potentially inappropriate prescribing identified through the Screening Tool of Older Persons' Prescriptions (STOPP) | From baseline to date of discharge from hospital, assessed up to 12 months
Change in potentially inappropriate prescribing identified through the Screening Tool of Older Persons' Prescriptions (STOPP) | From baseline to 12 months after discharge from hospital
Changes in medication, identified through screening of drug lists at their primary care physician. | 12 months after discharge from index hospital stay
  Drug changes made during hospitalization implemented by the primary care physician.
Changes in medication, identified through screening of drug lists at their primary care physician. | 3 months after discharge from index hospital stay
  Drug changes made during hospitalization implemented by the primary care physician.
Rehospitalizations where the reason for hospitalization is possibly, probably or certainly drug-related. | First rehospitalization after discharge from index hospital stay, up to 12 months after inclusion in study
  A chart review will be done retrospectively to evaluate if the patients first rehospitalization was drug related or not. Classified by a multiprofessional team of experts
Hip fracture | 12 months after discharge from index hospital stay
  Rate of hip fractures
Stroke | 12 months after discharge from index hospital stay
  Stroke rate during 12 months follow-up
The proportion of patients readmitted acutely within 30 days | 30 days after discharge from index hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Beate H Garcia, PhD, Principal Investigator — UiT The artic university of Norway
Locations (1):
- University hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansen JS, Havnes K, Halvorsen KH, Haustreis S, Skaue LW, Kamycheva E, Mathiesen L, Viktil KK, Granas AG, Garcia BH. Interdisciplinary collaboration across secondary and primary care to improve medication safety in the elderly (IMMENSE study): study protocol for a randomised controlled trial. BMJ Open. 2018 Jan 23;8(1):e020106. doi: 10.1136/bmjopen-2017-020106. PMID 29362276
- [Derived] Robinson EG, Gyllensten H, Granas AG, Halvorsen KH, Garcia BH. Health-related quality of life among older adults following acute hospitalization: longitudinal analysis of a randomized controlled trial. Qual Life Res. 2024 Aug;33(8):2219-2233. doi: 10.1007/s11136-024-03689-x. Epub 2024 Jun 17. PMID 38884880
- [Derived] Robinson EG, Gyllensten H, Johansen JS, Havnes K, Granas AG, Bergmo TS, Smabrekke L, Garcia BH, Halvorsen KH. A Trial-Based Cost-Utility Analysis of a Medication Optimization Intervention Versus Standard Care in Older Adults. Drugs Aging. 2023 Dec;40(12):1143-1155. doi: 10.1007/s40266-023-01077-7. Epub 2023 Nov 22. PMID 37991657
- [Derived] Johansen JS, Halvorsen KH, Svendsen K, Havnes K, Robinson EG, Wetting HL, Haustreis S, Smabrekke L, Kamycheva E, Garcia BH. Interdisciplinary collaboration across secondary and primary care to improve medication safety in the elderly (The IMMENSE study) - a randomized controlled trial. BMC Health Serv Res. 2022 Oct 26;22(1):1290. doi: 10.1186/s12913-022-08648-1. PMID 36289541